CLINICAL TRIAL: NCT00706316
Title: A Phase I Trial Evaluating the Administration of Epstein Barr Virus (EBV)-Specific Cytotoxic T-Lymphocytes (CTLs) to Patients With Recurrent or Metastatic EBV-Positive Nasopharygneal Cancer (NPC)
Brief Title: Administration of Epstein Barr Virus - Specific Cytotoxic T-Lymphocytes to Metastatic EBV-Positive Nasopharygneal Cancer
Acronym: NPC-CTL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: NPC-CTL
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Nasopharyngeal Cancer
Keywords: Nasopharygneal Cancer; Epstein Barr Virus; (EBV)-Specific Cytotoxic T-Lymphocytes; Recurrent; Metastatic; EBV-Positive Nasopharygneal Cancer
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Epstein-Barr Virus Infections; Recurrence; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EBV-Specific CTLs and CD45 Mab (Experimental): A dose escalation schema will be employed. Three to six patients will be treated at each of the following dose levels with EBV-Specific CTLs and CD45 Mab: Dose Level I: 2 x 10^7 cells/m2. Dose Level II: 5 x 10^7 cells/m2. Dose Level III: 1 x 10^8 cells/m2. Dose escalation decisions will be made after review of the data from the current dose level. There will be no intra-patient escalation. An additional 6-10 patients with measurable disease will be treated at the recommended phase II dose to expand the experience at this dose level.
  Interventions: Biological: EBV-Specific CTLs and CD45 Mab

INTERVENTIONS:
Biological: EBV-Specific CTLs and CD45 Mab — One time infusion (IV) at one of the following dose levels:
  Dose level I: 5 x 107 cells/m2
  Dose level II: 1 x 108 cells/m2
  Dose level III: 2 x 108 cells/m2

SUMMARY:
Nasopharyngeal cancer (NPC) is a cancer that starts at the back of the nose. Without distant spread, NPC is sensitive to radiotherapy and chemotherapy; however, if NPC relapses or spreads to other organs, treatment options are limited. This grant proposes to evaluate the safety and tolerability of a novel treatment for patients with NPC that has either relapsed or spread to distant organs. Epstein-Barr Virus (EBV) is known to play a role in the development of NPC, and studies have shown that NPC tumor cells express proteins that are related to EBV. Some of these proteins can trigger a response from the immune system, specifically the activation of cytotoxic T lymphocytes (CTLs), a type of immune cell that might exert anti-tumor effects. In this project, we will take blood from NPC patients, generate CTLs targeted against EBV, and re-infuse these back into patients in an attempt to achieve anti-tumor activity. Patients will also receive an antibody called CD45 Mab prior to CTL infusion in order to allow for better expansion of the infused CTLs in the patients.

DETAILED DESCRIPTION:
Nasopharyngeal cancer (NPC) is a cancer that starts at the back of the nose. Without distant spread, NPC is sensitive to radiotherapy and chemotherapy. However, the treatment of this cancer can lead to later complications, including other cancers, and if NPC relapses or spreads to other organs, the treatment options are limited. This grant proposes to evaluate the safety and tolerability of a novel treatment for patients with NPC that has either relapsed or spread to distant organs.

Epstein-Barr Virus (EBV) is known to play a role in the development of NPC in individuals, especially those with a compromised immune system. Studies have shown that NPC tumor cells express proteins that are related to EBV. Some of these proteins can trigger a response from the immune system, specifically the activation of cytotoxic T lymphocytes (CTLs), a type of immune cell that might exert anti-tumor effects. In this project, we will take blood from NPC patients, generate CTLs targeted against EBV, and re-infuse these back into patients in an attempt to achieve anti-tumor activity. Patients will also receive an antibody called CD45 Mab prior to CTL infusion in order to allow for better expansion of the infused CTLs in the patients.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with EBV positive NPC, with recurrent and/or metastatic disease
* Patients with a life expectancy > 3 months.
* Patients with an ECOG performance status of 0, 1 or 2
* No severe intercurrent infection.
* Patients who are able to give informed consent.
* Patients with:

  * bilirubin <2x normal,
  * SGOT (AST) and SGPT (ALT) <3x normal,
  * Hgb >80 g/L,
  * absolute neutrophil count (ANC) > 1.5 x 109/L,
  * and platelets > 100 x 109/L.
* Patients with a creatinine <2x normal for age
* Patients should have been off any chemotherapy or other investigational therapy for at least 4 weeks prior to entry in this study.
* Patients should have completed any prior radiation therapy for at least 3 weeks prior to entry in this study. Exception may be made, however, for low-dose, non-myelosuppressive radiotherapy, but this must be discussed with Principal Investigator(s).
* All patients must have measurable disease, with minimum indicator lesions size as follows:

  * CT scan > 2 cm (or > 1 cm if spiral CT scan is used)
  * Ultrasound > 2 cm
  * Chest x-ray > 2 cm
  * Physical exam > 1 cm (skin lesions, nodes, soft tissue masses)

Exclusion Criteria:

* Patients with a life expectancy of < 3 months.
* Patients with an ECOG performance status of >2.
* Patients with a severe intercurrent infection.
* Patients unable or unwilling to give informed consent.
* Patients with a bilirubin >2x normal.
* SGOT (AST) and SGPT (ALT) >3x normal.
* Patients with a creatinine >2x normal for age
* Patients with Hgb < 80 g/L, absolute neutrophil count (ANC) < 1.5 x 109/L, and platelets < 100 x 109/L.
* Due to unknown effects of this therapy on a fetus, pregnant women are excluded from this research. Lactating women are excluded from this study. Patients and their partners must use an effective birth control method during the study and for 6 months after. Effective birth control methods are: total abstinence, oral contraceptives, intrauterine devices, contraceptive implants under the skin or contraceptive injections. If one of these methods cannot be used, contraceptive foam with a condom is allowed. The male partner should use a condom.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-12; Primary Completion 2009-08 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
To determine the safety of autologous EBV-specific CTLs in patients with nasopharyngeal cancer | 24 months

SECONDARY OUTCOMES:
To obtain information on the expansion, persistence and anti-tumor effects of EBV-specific CTL lines in patients with nasopharyngeal cancer | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Siu, MD, Principal Investigator — University Health Network - Princess Margaret Hospital
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada